CLINICAL TRIAL: NCT03488524
Title: Evaluation of the Safety, Tolerability, Efficacy, and Activity of AMX0035, a Fixed Combination of Phenylbutyrate (PB) and Tauroursodeoxycholic Acid (TUDCA), for Treatment of Amyotrophic Lateral Sclerosis: Open-Label Extension
Brief Title: Open Label Extension Study of AMX0035 in Patients With ALS
Acronym: CENTAUR-OLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMX-3500-OLE
Record Dates: First submitted 2018-03-23; First posted 2018-04-05 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — sodium phenylbutyrate and taurursodiol; 4-phenylbutyric acid; ursodoxicoltaurine

STUDY DESIGN:
Intervention Model Description: This is an open-label extension study to CENTAUR (AMX3500)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMX0035 (Experimental): AMX0035 twice daily--a combination of Sodium Phenylbutyrate (3g) and Taurursodiol (1g)
  Interventions: Drug: AMX0035

INTERVENTIONS:
Drug: AMX0035 — Combination therapy of PB and TURSO
  Other Names: Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO, also known as Ursodoxicoltaurine or Tauroursodeoxycholic Acid [TUDCA])

SUMMARY:
This extension study, in which all participants received active treatment (AMX0035), was designed to assess the longer-term safety and therapeutic potential of AMX0035 for participants who have completed the Main Study (AMX3500, also known as CENTAUR).

DETAILED DESCRIPTION:
The Centaur Open Label Extension Study (CENTAUR-OLE) is an extension study for patients with ALS who participated in the CENTAUR study (Study AMX3500). During the OLE, all participants received active treatment (AMX0035), and the investigators, evaluators, and participants remained blinded to the randomized treatment assigned at the beginning of the double-blind main study. The study was designed to assess the longer term safety and therapeutic potential of AMX0035.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of all visits in the randomized, double blind AMX3500 study. Participants who received tracheostomy or permanent assisted ventilation (PAV) during the course of the main study could enroll in the OLE if they completed all visits in the main study.
2. Must enroll in the OLE within 28 days of the Week 24 visit of the main study.
3. Signed informed consent to enter the OLE phase.

Exclusion Criteria:

1. Discontinued study drug prematurely in the double-blind phase of the study for reasons other than tracheostomy or PAV.
2. Exposure to or anticipated requirement for any disallowed medication listed in the protocol.
3. Any ongoing adverse events that in the opinion of the Site Investigator are clear contraindications to the study drug.
4. Unstable cardiac or other life-threatening disease emergent during the randomized, double blind study
5. Any major medical condition that in the opinion of the Site Investigator would interfere with the study and place the subject at increased risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Paganoni, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (24):
- United States (24):
  - Barrow Neurological Institute-Dignity Health, St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, Irvine, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - University of Florida College of Medicine, Gainesville, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa, Carver College of Medicine, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Ochsner Neuroscience Institute, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Neurology Associates, PC, Lincoln, Nebraska
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Penn Comprehensive Neuroscience Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Neurology, PA, Dallas, Texas
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas
  - Swedish Neuroscience Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paganoni S, Watkins C, Cawson M, Hendrix S, Dickson SP, Knowlton N, Timmons J, Manuel M, Cudkowicz M. Survival analyses from the CENTAUR trial in amyotrophic lateral sclerosis: Evaluating the impact of treatment crossover on outcomes. Muscle Nerve. 2022 Aug;66(2):136-141. doi: 10.1002/mus.27569. Epub 2022 May 31. PMID 35508892
- [Result] Paganoni S, Hendrix S, Dickson SP, Knowlton N, Berry JD, Elliott MA, Maiser S, Karam C, Caress JB, Owegi MA, Quick A, Wymer J, Goutman SA, Heitzman D, Heiman-Patterson TD, Jackson C, Quinn C, Rothstein JD, Kasarskis EJ, Katz J, Jenkins L, Ladha SS, Miller TM, Scelsa SN, Vu TH, Fournier C, Johnson KM, Swenson A, Goyal N, Pattee GL, Babu S, Chase M, Dagostino D, Hall M, Kittle G, Eydinov M, Ostrow J, Pothier L, Randall R, Shefner JM, Sherman AV, Tustison E, Vigneswaran P, Yu H, Cohen J, Klee J, Tanzi R, Gilbert W, Yeramian P, Cudkowicz M. Effect of sodium phenylbutyrate/taurursodiol on tracheostomy/ventilation-free survival and hospitalisation in amyotrophic lateral sclerosis: long-term results from the CENTAUR trial. J Neurol Neurosurg Psychiatry. 2022 May 16;93(8):871-5. doi: 10.1136/jnnp-2022-329024. Online ahead of print. PMID 35577511
- [Result] Paganoni S, Hendrix S, Dickson SP, Knowlton N, Macklin EA, Berry JD, Elliott MA, Maiser S, Karam C, Caress JB, Owegi MA, Quick A, Wymer J, Goutman SA, Heitzman D, Heiman-Patterson TD, Jackson CE, Quinn C, Rothstein JD, Kasarskis EJ, Katz J, Jenkins L, Ladha S, Miller TM, Scelsa SN, Vu TH, Fournier CN, Glass JD, Johnson KM, Swenson A, Goyal NA, Pattee GL, Andres PL, Babu S, Chase M, Dagostino D, Hall M, Kittle G, Eydinov M, McGovern M, Ostrow J, Pothier L, Randall R, Shefner JM, Sherman AV, St Pierre ME, Tustison E, Vigneswaran P, Walker J, Yu H, Chan J, Wittes J, Yu ZF, Cohen J, Klee J, Leslie K, Tanzi RE, Gilbert W, Yeramian PD, Schoenfeld D, Cudkowicz ME. Long-term survival of participants in the CENTAUR trial of sodium phenylbutyrate-taurursodiol in amyotrophic lateral sclerosis. Muscle Nerve. 2021 Jan;63(1):31-39. doi: 10.1002/mus.27091. Epub 2020 Oct 30. PMID 33063909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the 24-week double-blind main study (Study AMX3500) on treatment were eligible to enter into the OLE.
Pre-assignment Details: To maintain the study blind, participants who entered the OLE initiated dosing in the OLE with 2 sachets of AMX0035 daily (ie, participants who switched from placebo to AMX0035 were not titrated using a starting dose of 1 sachet daily for the first 3 weeks, which was the starting dosing in the Main Study AMX3500).
Groups:
- AMX0035: AMX0035 twice daily--a combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO)
Period: Overall Study
Arm/Group | AMX0035
Started | 90
Completed | 2
Not Completed | 88
Not completed — Withdrawal by Subject | 51
Not completed — Death | 19
Not completed — Study Sponsor | 11
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Participants from the Main Study (AMX3500) who participated in the OLE study. Demographic and baseline characteristics for the Main Study can be found in record NCT03127514.
Groups:
- Placebo in Main Study-AMX0035 in OLE; AMX0035 in Main Study-AMX0035 in OLE: AMX0035 twice daily--a combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO)
- Total: Total of all reporting groups
Arm/Group | Placebo in Main Study-AMX0035 in OLE | AMX0035 in Main Study-AMX0035 in OLE | Total
Number analyzed (Participants) | 34 | 56 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (7.41) | 57.8 (10.22) | 58.0 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 24 | 43 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 33 | 52 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 33 | 52 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (6.50) | 26.8 (4.67) | 26.9 (5.40)
Del-FS: Rate of disease progression prior to entering the study [Mean (Standard Deviation); unit: ScaleScore/Months post-symptom onset] — DEL-FS score has been shown to be a strong predictor of functional decline. The score is calculated as the points lost on the ALSFRS-R from a maximum score of 48 divided by the months since symptom onset at baseline. Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available.
  ScaleScore/Months post-symptom onset
    number analyzed (Participants) | 32 | 54 | 86
    (all) | 1.03 (0.73) | 0.92 (0.46) | 0.96 (0.57)
Time since ALS diagnosis [Mean (Standard Deviation); unit: months] — Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available.
  months
    number analyzed (Participants) | 32 | 54 | 86
    (all) | 11.9 (3.54) | 11.7 (3.80) | 11.8 (3.69)
Time since onset of ALS symptoms [Mean (Standard Deviation); unit: months] — Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available.
  months
    number analyzed (Participants) | 32 | 54 | 86
    (all) | 19.2 (3.72) | 19.4 (4.29) | 19.3 (4.07)
Use of either edaravone or riluzole at or prior to study entry [Count of Participants; unit: Participants] — Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available.
  Participants
    number analyzed (Participants) | 32 | 54 | 86
    (all) | 28 | 45 | 73
Slow vital capacity (SVC) - % Predicted [Mean (Standard Deviation); unit: percent of predicted] — SVC volumes were standardized to predicted percent normalized values based on age, sex, and height. Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available. Not all participants had baseline data for this measure.
  percent of predicted
    number analyzed (Participants) | 29 | 53 | 82
    (all) | 72.7 (21.22) | 71.2 (23.12) | 71.7 (22.34)
ALS Functional Rating Scale - Revised (ALSFRS-R) total score [Mean (Standard Deviation); unit: scores on a scale] — The ALSFRS questionnaire is designed to determine the participant's assessment of their capability and independence in 12 functional activities relevant to ALS. ALSFRS-R consists of 12 items across 4 subdomains of function (bulbar, fine motor, gross motor, and breathing) with each item scored on a scale from 0 (total loss of function) to 4 (no loss of function). Total scores range from 0 to 48, with higher scores indicating better function. Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available.
  scores on a scale
    number analyzed (Participants) | 32 | 54 | 86
    (all) | 29.8 (9.36) | 30.6 (8.42) | 30.3 (8.74)
Accurate Test of Limb Isometric Strength (ATLIS) upper extremity score [Mean (Standard Deviation); unit: percent of predicted normal values] — The ATLIS device measures isometric strength in 6 upper extremity muscle groups (right and left grip strength, elbow extension and flexion). Raw values were standardized to percent predicted normal values for strength based on sex, age, weight, and height. Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available. Not all participants had baseline data for this measure.
  percent of predicted normal values
    number analyzed (Participants) | 28 | 45 | 73
    (all) | 43.29 (23.24) | 39.91 (23.74) | 41.21 (23.45)
Accurate Test of Limb Isometric Strength (ATLIS) lower extremity score [Mean (Standard Deviation); unit: percent of predicted normal values] — The ATLIS device measures isometric strength in 6 lower extremity muscle groups (left knee extension, right knee extension, left knee flexion, right knee flexion, left ankle dorsiflexion, right ankle dorsiflexion). Raw values were standardized to percent predicted normal values for strength based on sex, age, weight, and height. Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available. Not all participants had baseline data for this measure.
  percent of predicted normal values
    number analyzed (Participants) | 28 | 45 | 73
    (all) | 51.89 (25.22) | 49.98 (22.52) | 50.72 (23.45)
Accurate Test of Limb Isometric Strength (ATLIS) total score [Mean (Standard Deviation); unit: percent of predicted normal values] — The ATLIS device measures isometric strength in 6 lower extremity and 6 upper extremity muscle groups. Raw values were standardized to percent predicted normal values for strength based on sex, age, weight, and height. Population: Population for this measure is the mITT population, which included included all participants who received at least 1 dose of study medication in the main study who had at least 1 post baseline total ALSFRS-R score available. Not all participants had baseline data for this measure.
  percent of predicted normal values
    number analyzed (Participants) | 28 | 45 | 73
    (all) | 43.21 (23.20) | 39.82 (23.69) | 41.12 (23.40)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs from baseline in the OLE study through the last participant's last visit in the OLE
Time Frame: From the Baseline Visit in the OLE study through Week 132 or the Early Discontinuation (Final Safety) Visit for each participant (for up to approximately 132 weeks)
Population: Safety Population, which included all participants who received at least 1 dose of study medication in the OLE.
Measure: Count of Participants; unit: Participants
Groups:
- AMX0035 in OLE: AMX0035 twice daily--a combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO)
Arm/Group | AMX0035 in OLE
Number analyzed (Participants) | 90
Participants | 81

2. Secondary Outcome: Amyotrophic Lateral Sclerosis Rating Scale Revised Total Score (ALSFRS-R) Change in Slope
Description: Comparison of the difference in change in slope of Amyotrophic Lateral Sclerosis Rating Scale Revised (ALSFRS-R) total score from the Main Study baseline through Week 48 of the open-label extension (OLE) between the 2 treatment groups: those randomized to AMX0035 in the Main Study and those randomized to Placebo in the main study (all participants in the OLE received AMX0035). The slope is measured as a change in score divided by a change in time. ALSFRS-R consists of 12 items across 4 subdomains of function (bulbar, fine motor, gross motor, and breathing) with each item scored on a scale from 0 (total loss of function) to 4 (no loss of function). Total scores range from 0 to 48, with higher scores indicating better function.
Time Frame: From baseline in the Main Study through Week 24 of the OLE (48 weeks overall)
Population: mITT Population. Participants from the Main Study who did not enter the OLE were included.
Measure: Least Squares Mean (Standard Error); unit: Change in ALSFRS-R Total Score per Month
Groups:
- Randomized to Placebo in Main Study and Did or Did Not Participate in OLE; Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE: AMX0035 twice daily--a combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO)
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 87
Change in ALSFRS-R Total Score per Month | 17.38 (1.545) | 21.61 (1.178)
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Participants who did not enter the open-label extension (OLE) were included in this analysis; Test type: Superiority; p = 0.0239, Mixed Models Analysis — Significance testing was 2-tailed and considered statistically significant if the calculated p-value was ≤0.05; Random-slope, shared-baseline, linear mixed model was adjusted for age and prebaseline ALSFRS-R slope; Mean Difference (Final Values) = 4.23, 95% CI 2-sided [0.56 to 7.90], Standard Error of Mean 1.870

3. Secondary Outcome: Survival - Time to Death
Description: Median survival in months
Time Frame: From date of first dose in the Main Study (each participant's Baseline Visit) through up to approximately 42 months (approximately 182 weeks)
Population: ITT Population. Participants from the Main Study who did not enter the OLE were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 89
Months | 18.7 [13.5 to 24.4] | 23.5 [19.5 to 26.2]
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Cox Proportional Hazards analysis; Test type: Superiority; p = 0.0475, Hazard ratio; Hazard Ratio (HR) = 0.644, 95% CI 2-sided [0.416 to 0.995]

4. Secondary Outcome: Composite of Time to Hospitalization, Death or Death Equivalent
Description: The composite endpoint of time to hospitalization, death or death equivalent was defined as hospitalization, death, tracheostomy or PAV. PAV is defined as more than 22 hours daily of non-invasive mechanical ventilation for more than 1 week (7 days).
Time Frame: as for outcome 3
Population: ITT population. Participants from the Main Study who did not enter the OLE were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 89
Months | 10.0 [6.1 to 12.7] | 14.8 [10.7 to 18.2]
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Test type: Superiority; p = 0.0308, Hazard Ratio; Hazard Ratio (HR) = 0.621, 95% CI 2-sided [0.403 to 0.957]

5. Secondary Outcome: Accurate Testing of Limb Isometric Strength (ATLIS) Change in Slope - Upper Extremities
Description: Comparison of the difference in change in slope of Accurate Testing of Limb Isometric Strength (ATLIS) upper extremity score from the Main Study baseline through Week 48 of the open-label extension (OLE) between the 2 treatment groups: those randomized to AMX0035 in the Main Study and those randomized to Placebo in the main study (all participants in the OLE received AMX0035). The ATLIS device measures isometric strength in 6 upper extremity muscle groups. Raw values were standardized to percent predicted normal values for strength based on sex, age, weight, and height.
Time Frame: From baseline in the Main Study through Week 24 of the OLE (48 weeks overall)
Population: mITT Population. Participants from the Main Study who did not enter the OLE were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: % of Predicted Normal Change per Month
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 87
% of Predicted Normal Change per Month | 12.06 (3.283) | 19.83 (2.591)
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Test type: Superiority; p = 0.0291, Mixed Models Analysis; Mean Difference (Final Values) = 7.77, 95% CI 2-sided [0.80 to 14.75], Standard Error of Mean 3.550

6. Secondary Outcome: Accurate Testing of Limb Isometric Strength (ATLIS) Change in Slope - Lower Extremities
Description: Comparison of the difference in change in slope of Accurate Testing of Limb Isometric Strength (ATLIS) lower extremity score from the Main Study baseline through Week 48 of the open-label extension (OLE) between the 2 treatment groups: those randomized to AMX0035 in the Main Study and those randomized to Placebo in the main study (all participants in the OLE received AMX0035). The ATLIS device measures isometric strength in 6 lower extremity muscle groups. Raw values were standardized to percent predicted normal values for strength based on sex, age, weight, and height.
Time Frame: From baseline in the Main Study through Week 24 of the OLE (48 weeks overall)
Population: mITT Population. Participants from the Main Study who did not enter the OLE were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: % of Predicted Normal Change per Month
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 87
% of Predicted Normal Change per Month | 20.48 (3.653) | 25.24 (2.893)
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Test type: Superiority; p = 0.2261, Mixed Models Analysis; Mean Difference (Final Values) = 4.76, 95% CI 2-sided [-2.95 to 12.47], Standard Error of Mean 3.923

7. Secondary Outcome: Slow Vital Capacity Change in Slope
Description: Comparison of the difference in change in slope of Slow Vital Capacity (SVC) from the Main Study baseline through Week 48 of the open-label extension (OLE) between the 2 treatment groups: those randomized to AMX0035 in the Main Study and those randomized to Placebo in the main study (all participants in the OLE received AMX0035). SVC volumes were standardized to predicted percent normalized values for respiratory muscle function based on age, sex, and height.
Time Frame: From baseline in the Main Study through Week 24 of the OLE (48 weeks overall)
Population: mITT Population. Participants from the Main Study who did not enroll in the OLE were included.
Measure: Least Squares Mean (Standard Error); unit: % of Predicted Normal Change per Month
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 87
% of Predicted Normal Change per Month | 37.85 (4.427) | 48.52 (3.356)
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Test type: Superiority; p = 0.0372, Mixed Models Analysis — Nominal p-value; Mean Difference (Final Values) = 10.66, 95% CI 2-sided [0.63 to 20.69], Standard Error of Mean 5.103

8. Secondary Outcome: Accurate Testing of Limb Isometric Strength (ATLIS) Total Score Change in Slope
Description: Comparison of the difference in change in slope of Accurate Testing of Limb Isometric Strength (ATLIS) total score from the Main Study baseline through Week 48 of the open-label extension (OLE) between the 2 treatment groups: those randomized to AMX0035 in the Main Study and those randomized to Placebo in the main study (all participants in the OLE received AMX0035). The ATLIS device measures isometric strength in 6 upper and 6 lower extremity muscle groups. Raw values were standardized to percent predicted normal values for strength based on sex, age, weight, and height.
Time Frame: From Baseline in the Main Study through Week 24 in the OLE (48 weeks overall)
Population: mITT Population. Participants from the Main Study who did not enter the OLE were included.
Measure: Least Squares Mean (Standard Error); unit: % of Predicted normal change per month
Arm/Group | Randomized to Placebo in Main Study and Did or Did Not Participate in OLE | Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE
Number analyzed (Participants) | 48 | 87
% of Predicted normal change per month | 16.65 (2.973) | 22.84 (2.371)
Statistical Analysis 1: Comparison: Randomized to Placebo in Main Study and Did or Did Not Participate in OLE vs Randomized to AMX0035 in Main Study and Did or Did Not Participate in OLE; Test type: Superiority; p = 0.0503, Mixed Models Analysis — Nominal p-value

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline in the OLE study through study completion (generally about 2.5 years). Vital status was collected from date of first dose in the Main Study (each participant's Baseline Visit) through up to approximately 42 months (approximately 182 weeks)
Description: Symptoms of progression/worsening of ALS, including 'normal' progression, were to be recorded as AEs.
Arm/Group | AMX0035
All-Cause Mortality (participants affected / at risk) | 19/90
Serious Adverse Events (participants affected / at risk) | 31/90
Other Adverse Events (participants affected / at risk) | 81/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMX0035 (N=90)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Catheter site infection (Infections and infestations) | 1
Diverticulits (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Medical device site infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Dysphagia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Device malfunction (Product Issues) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMX0035 (N=90)
Nausea (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Urinary tract infection (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 20
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Weight decreased (Investigations) | 6
Disease progression (General disorders) | 5
Pyrexia (General disorders) | 5
Anxiety (Psychiatric disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT03488524/Prot_000.pdf
  • Statistical Analysis Plan: Primary SAP (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT03488524/SAP_001.pdf
  • Statistical Analysis Plan: Integrated Survival Analysis SAP (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03488524/SAP_002.pdf
  • Statistical Analysis Plan: Addendum to Integrated Survival Analysis SAP (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT03488524/SAP_003.pdf